CLINICAL TRIAL: NCT06047405
Title: NIV for Hypercapnic Respiratory Failure: AVAPS vs S/T BIPAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0745
Record Dates: First submitted 2023-08-10; First posted 2023-09-21 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: AVAPS; BIPAP; Hypercapnic respiratory failure; Noninvasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients from medical ICU or telemetry units will be randomized to one of the following arms:
  Arm 1: AVAPS mode Arm 2: BIPAP S/T mode
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Average Volume-Assured Pressure Support (AVAPS) (Active Comparator): Average Volume-Assured Pressure Support (AVAPS) setting on the noninvasive ventilator. The exact AVAPS setting will be titrated by the clinical team involved directly in the patient's care based on patient comfort and clinical response.
  Interventions: Device: Average Volume-Assured Pressure Support (AVAPS)
- Bilevel Positive Airway Pressure Spontaneous Timed (BIPAP S/T) (Active Comparator): Bilevel Positive Airway Pressure Spontaneous Timed (BIPAP S/T) setting on the noninvasive ventilator. The exact BIPAP S/T setting will be titrated by the clinical team involved directly in the patient's care based on patient comfort and clinical response.
  Interventions: Device: Bilevel Positive Airway Pressure Spontaneous Timed (BIPAP S/T)

INTERVENTIONS:
Device: Average Volume-Assured Pressure Support (AVAPS) — A setting on noninvasive ventilator that allows setting of maximum and minimum inspiratory pressure and sets a target tidal volume. The inspiratory pressure varies breath to breath to ensure pre-set tidal volume is delivered.
  Arms: Average Volume-Assured Pressure Support (AVAPS)
Device: Bilevel Positive Airway Pressure Spontaneous Timed (BIPAP S/T) — A setting on noninvasive ventilator that allows setting of inspiratory pressure, inspiratory time, expiratory pressure, and backup rate to deliver variable tidal volumes.
  Arms: Bilevel Positive Airway Pressure Spontaneous Timed (BIPAP S/T)

SUMMARY:
The goal of this study is to compare two different modes of noninvasive ventilation in hypercapnic respiratory failure. The investigators will compare AVAPS and BIPAP S/T and hypothesize that AVAPS will result in a decreased length of stay in the ICU or on telemetry. Currently, noninvasive ventilation is the standard of care for hypercapnic respiratory failure. However, the most effective mode for patients with hypercapnic respiratory failure is unclear.

DETAILED DESCRIPTION:
1. Overall Study Design and Plan

This is a single center, randomized trial that will include a total of 100 adult subjects aged 18 or older with hypercapnic respiratory failure of all etiologies (i.e. "all comers"). The investigators will randomize patients in a single-blinded (patient blinded) fashion to BIPAP S/T or AVAPS during the duration of their hospitalization. The investigators will assess ABG at baseline, 1 hour after initial placement on BIPAP S/T or AVAPS, and between hours 24-48 of use. The investigators will record the pre-NIV pH and PaCO2, post-NIV pH and PaCO2, length of hospital stay in the medical ICU or telemetry unit, days on NIV, need for intubation (if occurred), transition to medical ICU care in patients who were initially admitted to telemetry, and in-hospital mortality. All collected laboratory data are already done as part of usual care for all patients placed on NIV when a patient is on the telemetry unit or medical ICU. The groups will undergo stratified randomization based on whether they are initially admitted to medical ICU or medical telemetry. Patients from medical ICU or telemetry units will be randomized to one of the following arms:

Arm 1: AVAPS mode Arm 2 2: BIPAP S/T mode

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form directly by the patient; consent can also be obtained via a legal patient representative/health care proxy/surrogate
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older
4. Diagnosed with hypercapnic respiratory failure on admission (ABG)
5. Admitted to Lenox Hill Hospital medical intensive care unit or telemetry unit
6. Requiring noninvasive ventilation as determined by the treating physician for the treatment of hypercarbic respiratory failure

Exclusion Criteria:

1. Patients who require ventilation at predetermined tidal volumes
2. Patients who require rapid and frequent IPAP adjustments to maintain a consistent tidal volume
3. Age less than 18 years of age
4. Currently intubated
5. Chronic tracheostomy
6. Pregnancy
7. Hypotension
8. Epistaxis (nosebleed)
9. Untreated pertussis
10. Acute sinusitis or Otitis media
11. Patients at risk of aspirating gastric contents
12. Patients with lack of spontaneous respiratory drive
13. Patients with the inability to maintain a patent airway or adequately clear secretions
14. Prisoners or other institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay of telemetry length of stay | within one week of hospital discharge (5-7 days)
  In patients admitted to the medical ICU, the primary endpoint is ICU length of stay. This will be the number of days a patient is admitted from day 1 of admission until the day of discharge. In patients admitted to medical telemetry unit, the outcome is telemetry length of stay. This will be the number of days a patient is admitted from day 1 of admission until the day of discharge.

SECONDARY OUTCOMES:
Difference in PaCO2 value with NIV | within 24-48 hours after noninvasive ventilation
  Change in paCO2 on ABG (paCO2 before and after NIV use, measured as a numerical value in mmHg)
Time to normalization of pH | at the time of hospital discharge (an average of 5-7 days)
  Time to normalization of pH (hours)
Normalization of pH | at the time of hospital discharge (an average of 5-7 days)
  Return to normal range of pH as defined by the laboratory normal values (Binary measure)
Days on NIV | within one week of hospital discharge (5-7 days)
  Days on noninvasive ventilation
Need for intubation | within one week of hospital discharge (5-7 days)
  Need for intubation
Need for ICU stay | within one week of hospital discharge (5-7 days)
  Need for ICU stay (if disposition changed from telemetry unit)
Subgroup analysis (logistic regression or p-value) comparing outcomes 1- ICU or telemetry length of stay based on the underlying cause of hypercapnic respiratory failure | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for these outcome- for 1. ICU or telemetry length of stay. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.
Subgroup analysis (logistic regression or p-value) comparing outcome 2- difference in paCO2 reported as difference between groups (with p-value and/or standard deviation) | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for outcome 2- difference in PaCO2. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.
Subgroup analysis (logistic regression or p-value) comparing outcome 4- time to normalization of pH reported as difference between groups (with p-value and/or standard deviation) | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for outcome 4- time to normalization of pH. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.
Subgroup analysis (logistic regression or p-value) comparing outcome 5- days on NIV reported as difference between groups (with p-value and/or standard deviation) | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for outcome 5- days on NIV. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.
Subgroup analysis (logistic regression or p-value) comparing outcome 6- need for intubation reported as difference between groups (with p-value and/or standard deviation) | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for outcome 6- need for intubation. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.
Subgroup analysis (logistic regression or p-value) comparing outcome 7- need for ICU stay reported as difference between groups (with p-value and/or standard deviation) | through study completion, an average of 1 year
  We will perform subgroup analysis of each cause of hypercapnic respiratory failure (such as COPD, pulmonary edema, altered mental status, etc) for outcome 7- need for ICU stay. We will use either logistic regression model or p-value to determine the difference for each subgroup. The results will be reported as difference between groups with statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Oks, MD, Principal Investigator — Lenox Hill Hospital/Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only researchers on involved in conducting the study will have access to the information collected in the study.
  9.3 Data Handling and Record Keeping 9.3.1 Data Collection and Management All information accessed from the medical record will be de-identified. All data will be stored on an encrypted secure server, REDCap.
  9.3.2 Confidentiality and Privacy Privacy will be protected as data will be collected within the Northwell Redcap data portal. All data will be de-identified prior to entry into REDCap. All communication between subjects and researchers will be conducted in a private setting.

REFERENCES:
- [Background] Briones-Claudett KH, Esquinas Rodriguez A, Briones-Claudett MH, Puga-Tejada M, Cabrera Banos MDP, Pazmino Duenas CR, Torres Herrera CI, Grunauer M. Use of noninvasive mechanical ventilation with pressure support guaranteed with average volume in de novo hypoxaemic respiratory failure. A pilot study. Anaesthesiol Intensive Ther. 2018;50(4):283-290. doi: 10.5603/AIT.a2018.0036. Epub 2018 Oct 14. PMID 30317536
- [Background] Patout M, Gagnadoux F, Rabec C, Trzepizur W, Georges M, Perrin C, Tamisier R, Pepin JL, Llontop C, Attali V, Goutorbe F, Pontier-Marchandise S, Cervantes P, Bironneau V, Portmann A, Delrieu J, Cuvelier A, Muir JF. AVAPS-AE versus ST mode: A randomized controlled trial in patients with obesity hypoventilation syndrome. Respirology. 2020 Oct;25(10):1073-1081. doi: 10.1111/resp.13784. Epub 2020 Feb 13. PMID 32052923
- [Background] Magdy DM, Metwally A. Effect of average volume-assured pressure support treatment on health-related quality of life in COPD patients with chronic hypercapnic respiratory failure: a randomized trial. Respir Res. 2020 Mar 6;21(1):64. doi: 10.1186/s12931-020-1320-7. PMID 32143652
- [Background] Crisafulli E, Manni G, Kidonias M, Trianni L, Clini EM. Subjective sleep quality during average volume assured pressure support (AVAPS) ventilation in patients with hypercapnic COPD: a physiological pilot study. Lung. 2009 Sep-Oct;187(5):299-305. doi: 10.1007/s00408-009-9167-1. Epub 2009 Aug 13. PMID 19672655
- [Background] Storre JH, Seuthe B, Fiechter R, Milioglou S, Dreher M, Sorichter S, Windisch W. Average volume-assured pressure support in obesity hypoventilation: A randomized crossover trial. Chest. 2006 Sep;130(3):815-21. doi: 10.1378/chest.130.3.815. PMID 16963680
- [Background] Rose L, Hawkins M. Airway pressure release ventilation and biphasic positive airway pressure: a systematic review of definitional criteria. Intensive Care Med. 2008 Oct;34(10):1766-73. doi: 10.1007/s00134-008-1216-3. Epub 2008 Jul 17. PMID 18633595
- [Result] Goren NZ, Sanci E, Ercan Coskun FF, Gursoylu D, Bayram B. Comparison of BPAP S/T and Average Volume-Assured Pressure Support Modes for Hypercapnic Respiratory Failure in the Emergency Department: A Randomized Controlled Trial. Balkan Med J. 2021 Sep;38(5):265-271. doi: 10.5152/balkanmedj.2021.20137. PMID 34462252
- [Result] Briones Claudett KH, Briones Claudett M, Chung Sang Wong M, Nuques Martinez A, Soto Espinoza R, Montalvo M, Esquinas Rodriguez A, Gonzalez Diaz G, Grunauer Andrade M. Noninvasive mechanical ventilation with average volume assured pressure support (AVAPS) in patients with chronic obstructive pulmonary disease and hypercapnic encephalopathy. BMC Pulm Med. 2013 Mar 12;13:12. doi: 10.1186/1471-2466-13-12. PMID 23497021
- [Result] Murphy PB, Davidson C, Hind MD, Simonds A, Williams AJ, Hopkinson NS, Moxham J, Polkey M, Hart N. Volume targeted versus pressure support non-invasive ventilation in patients with super obesity and chronic respiratory failure: a randomised controlled trial. Thorax. 2012 Aug;67(8):727-34. doi: 10.1136/thoraxjnl-2011-201081. Epub 2012 Mar 1. PMID 22382596